CLINICAL TRIAL: NCT07175376
Title: Resilience Enhancement Utilizing an Electronic Frailty Index-Directed Care Pathway for Older Adults Receiving Chemotherapy (RESILIENCE-e): A Prospective Single-Arm Interventional Study
Brief Title: Resilience Enhancement Using Electronic Frailty Index-Directed Care Pathway
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Wake Forest Baptist (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00135936; ONC-CCS-2413 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Frail; Chemotherapy
Keywords: Cancer; Frailty Index; eFI score
MeSH Terms: conditions — Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants 65 years or older with active cancer diagnosis and planned chemotherapy (Experimental): Participants aged 65 or older with an active cancer diagnosis who are planned to receive chemotherapy and are eFI pre-frail or frail. Participants will be provided with results and education regarding baseline assessments and offered referrals for supportive care interventions to decrease chemotherapy toxicity
  Interventions: Other: Supportive Care

INTERVENTIONS:
Other: Supportive Care — Geriatric assessment (GA) -guided supportive care and weekly Patient Reported Outcomes (PRO) symptom assessment

SUMMARY:
The study purpose is to gain a better understanding of the needs of adults aged 65 and older while they are receiving chemotherapy by measuring their resilience and tailor care plans based on their individual needs.

DETAILED DESCRIPTION:
This is a prospective single-arm intervention trial of patients aged 65 or older with an active cancer diagnosis who are planned to receive chemotherapy and are eFI (Electronic Health Record (EHR)-based frailty index) pre-frail or frail.

Patients will be enrolled before initiation of chemotherapy. Following a baseline assessment, subjects will be provided with results regarding their frailty, will be offered referrals for supportive care interventions and will participate in weekly symptom reporting (electronic survey + phone call from research nurse) for 12 weeks. Follow-up assessments will be completed at 12 weeks and a subset of participants and providers in participating clinics will be contacted to consent and participate in an interview to provide feedback on the intervention including barriers/facilitators.

ELIGIBILITY:
Inclusion Criteria:

Patients with cancer:

* Ability to understand and willingness to sign an IRB-approved informed consent
* Age ≥ 65 years at the time of enrollment.
* Planned to initiate an outpatient chemotherapy regimen for cancer treatment (any type or stage), either as an initial therapy or as a new line of therapy, with curative or palliative intent.
* eFI pre-frail or frail status (available in EHR) within 30 days before enrollment.
* Ability to read and understand the English language

Providers:

* Treating medical oncologist of at least one patient participant who enrolled on to the study and completed baseline assessment.

Exclusion Criteria:

Patients:

* Documented physical or psychological comorbidity that would limit participant's ability to understand or comply with study procedures for the entire length of the study per the enrolling investigator.
* Chemotherapy planned at a facility outside the Atrium Health system.
* Currently receiving chemotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Enrollment
  The proportion of patients who are enrolled out of the total number of eligible patients approached for enrollment
Retention rate | At 12 weeks after initiation of standard of care chemotherapy
  The proportion of enrolled patient participants who complete Visit 2 out of the total number of patient participants who were enrolled and initiate chemotherapy
Completion rate of Weekly Symptom Assessment | Weeks 1 to 12
  The total number of weekly assessments completed out of the total number of weekly assessments among participants who enroll and initiate chemotherapy.

SECONDARY OUTCOMES:
Number of Participants with Hospital admission | Baseline to Week 12
  Number of participants with hospital admissions during the 12 weeks after chemotherapy initiation
Number of Participants with ED visits | Baseline to Week 12
  Number of participants with Emergency Department (ED) visits during the 12 weeks after chemotherapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No